CLINICAL TRIAL: NCT03915106
Title: Evaluation of Health-related Quality of Life (HRQoL) of Adolescent Idiopathic Scoliosis (AIS) Patients Who Require Bracing or Surgery Using SRS-22 Questionnaire
Brief Title: Quality of Life (HRQoL) of AIS Patients Who Require Bracing or Surgery Using SRS-22 Questionnaire
Acronym: QolAISSRS22
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Alec Lik-Hang Hung, Principal Investigator, Chinese University of Hong Kong
Other Study IDs: 2019.213
Record Dates: First submitted 2019-04-10; First posted 2019-04-16 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Scoliosis; Adolescence; Adolescent; Quality of Life; SRS
Keywords: scoliosis; adolescent idiopathic scoliosis; bracing; surgery; quality of life; questionnaire
MeSH Terms: conditions — Scoliosis | interventions — Braces

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Bracing: AIS patients undergoing bracing to control the spinal curve progression
  Interventions: Device: Brace
- Surgical: Severe AIS patients requiring surgical intervention to correct the spinal curve
  Interventions: Procedure: Surgical correction using implants

INTERVENTIONS:
Device: Brace — Wear a rigid brace
  Groups: Bracing
Procedure: Surgical correction using implants — Surgical correction of spine using implants (metallic rods and metallic screws)
  Groups: Surgical

SUMMARY:
Adolescent Idiopathic Scoliosis (AIS) is an unexpected curvature of spine at teenage. AIS causes mainly unpleasant appearance, and sometime comes with pain and difficult to locate or move around. When the spinal curve, or "Cobb angle", increases with time, the investigators call it severe condition when the Cobb angle is 60 degrees or above. The severe suffering patients need to be operated to correct their spinal curve by using metallic rods and metallic screws (implants) to fix the spine. In order to avoid this surgery, the investigators use "brace", a hard fitting case, trying to control the spinal curve degree by using forces from outside. (bracing) to intervene the spinal curve progression is highly recommended for patients with particular clinical characteristics. However, bracing is not always a present experience apart from function restriction. Clinical recommendation requires the patients to brace over 20 hours everyday, which means the patients have to be "braced" around the clock. Patients' perception on being "braced" all day, apart from discomforts under bracing, self-image and mental health after bracing are also important psycho-social factors which have yet to be addressed. Based on our clinical experience, 1-2% of AIS patients, undergoing bracing or not (i.e. at observation stage), require surgical intervention due to rapid spinal progression in a short period of time. By definition, surgery will be arranged for patients with major spinal curve ≥50. The use of health-related-quality-of-life (HRQoL) questionnaires allow clinical professionals to explore many different kinds of interests on patients, including the patient's feeling on his/her medical condition and satisfaction with provided care. Scoliosis Research Society (SRS) patient outcome tool has been a well-accepted HRQoL questionnaire to look for the perception of patients with spinal problems of their status. The SRS-22 questionnaire that has been well accepted as its trustworthy on the score results and SRS-22 is good to be used in patients under different conditions across the disease. This is very important to obtain and compare the scores over time in order to look for any consistent changes. Apart from AIS patients requiring bracing, surgical cases are also very important group of patients to monitor their quality of life before and after surgery, and every follow-up visit after surgery.

DETAILED DESCRIPTION:
Adolescent Idiopathic Scoliosis (AIS) is a 3D deformity of spine happened with unidentifiable cause at teenage. AIS causes mainly cosmetic problems with a lesser incidence of functional deficit and pain. AIS patients under severe condition, defined as the major spinal curve angle named "Cobb angle" larger than 60 degrees, requires surgical intervention to the spinal curve with implants permanently applied along the spine. The use of "brace" (bracing) to intervene the spinal curve progression is highly recommended for patients with particular clinical characteristics. However, bracing is not always a present experience apart from function restriction. Clinical recommendation requires the patients to brace over 20 hours everyday, which means the patients have to be "braced" around the clock. Patients' perception on being "braced" all day, apart from discomforts under bracing, self-image and mental health after bracing are also important psycho-social factors which have yet to be addressed. Based on our clinical experience, 1-2% of AIS patients, undergoing bracing or not (i.e. at observation stage), require surgical intervention due to rapid spinal progression in a short period of time. By definition, surgery will be arranged for patients with major spinal curve ≥50 degrees.

The health-related-quality-of-life (HRQoL) questionnaires allow clinical professionals to explore many areas of interest, including the patient's perception of his/her condition and satisfaction with provided care. Scoliosis Research Society (SRS) Outcomes Instrument has been an accepted HRQoL questionnaire to evaluate the perception of patients with spinal deformities of their status. The SRS-22 questionnaire that has been shown to have high reliability and concurrent validity and discrimination validity and responsiveness to change. SRS-22 questionnaire comprises 22 questions under 5 domains (function, pain, self-image, mental health, and satisfaction with management). Through these 22 questions, the psycho-social status can be quantified in terms of "scores" and the scores obtained at different time points can be compared. Continuous monitoring of these factors are important along the bracing period to look for patients with continuously poor psycho-social status of which bracing period is possibly last for years. Apart from AIS patients requiring bracing, surgical cases are also very important group of patients to monitor their quality of life before and after surgery, and every follow-up visit after surgery.

ELIGIBILITY:
Inclusion Criteria:

* AIS patients who attend the scoliosis clinic at specialized outpatient clinic in Prince of Wales hospital and require wearing brace, or patients who suffer from severe scoliosis and require surgery on their first clinic visit
* Can read and understand either English or Chinese

Exclusion Criteria:

* To observe (i.e. not require to wear brace) after clinic visit
* Cannot read or understand either English or Chinese

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients visiting a specialized clinic at Prince of Wales Hospital, Shatin, Hong Kong
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline SRS-22 Function score at 1 year | Baseline and 1 year
  Select 1 from 5 answers in each question. Scores from 1 to 5 (1, 2, 3, 4, and 5), the higher score the better outcome. A calculated score. "Function" score was calculated by adding the scores from questions 1 to 4.
Change from baseline SRS-22 Pain score at 1 year | Baseline and 1 year
  Select 1 from 5 answers in each question. Scores from 1 to 5 (1, 2, 3, 4, and 5), the higher score the better outcome. A calculated score. "Pain" score was calculated by adding the scores from questions 5 to 8.
Change from baseline SRS-22 Self-image score at 1 year | Baseline and 1 year
  Select 1 from 5 answers in each question. Scores from 1 to 5 (1, 2, 3, 4, and 5), the higher score the better outcome. A calculated score. "Self-image" score was calculated by adding the scores from questions 9 to 12.
Change from baseline SRS-22 Mental score at 1 year | Baseline and 1 year
  Select 1 from 5 answers in each question. Scores from 1 to 5 (1, 2, 3, 4, and 5), the higher score the better outcome. A calculated score. "Mental" score was calculated by adding the scores from questions 13 to 16.
Change from baseline SRS-22 Satisfaction score at 1 year | Baseline and 1 year
  Select 1 from 5 answers in each question. Scores from 1 to 5 (1, 2, 3, 4, and 5), the higher score the better outcome. A calculated score. "Satisfaction" score was calculated by adding the scores from questions 17 to 20.

CONTACTS AND LOCATIONS:
Overall Officials: Alec Lik-Hang Hung, Dr., Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No